CLINICAL TRIAL: NCT06647290
Title: Excision and Negative Pressure Wound Therapy Versus Excision and Leaving Open With Standard Wound Care for Management of Chronic Pilonidal Sinus Disease - A Randomised Controlled Trial
Brief Title: ENVELOP: Wound Care Following Pilonidal Sinus Surgery
Acronym: ENVELOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCSI-ENVELOP
Record Dates: First submitted 2023-11-28; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Pilonidal Sinus; Wound Healing
Keywords: Negative Pressure Wound Therapy; Surgical Site Infection; Post-operative Complications; Health Economics; POSAS; CoPaQ; EQ-5D-5L; Pain Score
MeSH Terms: conditions — Pilonidal Sinus; Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): The wound is dressed using negative pressure wound therapy.
  Interventions: Device: Negative Pressure Wound Therapy
- Standard Wound dressing (Active Comparator): After the skin is closed, the wound is covered using sterile standard gauze dressing.
  Interventions: Device: Negative Pressure Wound Therapy

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — Application of a negative wound pressure therapy dressing to the wound post laparotomy

SUMMARY:
This is a single-blinded, multicentre, prospective randomised controlled trial (RCT) comparing post-operative and patient-reported outcomes for patients undergoing application of negative-pressure wound therapy (NPWT) after sinus tract excision as compared to excision and standard open wound care in chronic pilonidal sinus disease (PSD).

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is a chronic inflammatory condition of the skin and subcutaneous tissues arising from hair follicles in the natal cleft. The definitive aetiology of the condition is unknown, however, it is theorised that it is the result of either the obstruction and subsequent inflammation of hair follicles or secondary to hair penetrating through the skin into the subcutaneous tissue. This results in infection, abscess formation, chronic discharge and pain. PSD is a common condition affecting 26 per 10,000 population, with the prevalence reaching 1.1% in young adult males.

PSD causes a significant burden on healthcare services due to high rates of recurrence and readmission following surgery, together with negative impacts on patients' quality of life and self-image. An effective management strategy for the disease is necessary to ensure that post-operative outcomes are optimised and patient-reported outcomes are satisfactory in those whose PSD requires surgery.

The objective of this multicentre, national RCT is to prospectively investigate the effect of negative pressure wound therapy compared to leaving open with standard wound care on time to wound healing following surgical excision of chronic PSD.

ELIGIBILITY:
Inclusion Criteria:

i) They are aged 18 years or older

ii) They are undergoing elective pilonidal sinus excision without primary closure

Exclusion Criteria:

i) They are unable to adhere to protocol requirements e.g. questionnaire completion

ii) They are undergoing emergency drainage for a pilonidal abscess

iii) They are undergoing surgery for a pilonidal sinus disease in locations other than the natal cleft

iv) They have underlying osteomyelitis

v) They have underlying fistulating disease e.g. Crohn's

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-27 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound healing | 6 months post surgery
  Number of days to complete epithelialisation or closure of the wound without any discharge, drainage, scab, and/or the requirement for further dressing. The quality of wound healing will be assessed using a validated patient and observer reported scar assessment tool-POSAS.

SECONDARY OUTCOMES:
Measure of post operative pain | 6 months post surgery
  Pain measured by visual analogue pain scores which is a scale from 1 (no pain) to 10 (worst pain), between the NPWT and SWC Groups.
Measure of post operative complications | 6 months post surgery
  Measure of post operative complications between the NPWT and SWC Groups
Measure of quality of life | 6 months post surgery
  To compare quality-of-life differences between the two groups from the time of surgery until wound healing is achieved using the
To investigate resource use | 6 months post surgery
  To investigate resource use and thereby cost effectiveness of NPWT versus standard wound care
To compare recurrence rates | 6 months post surgery
  To compare the 6-month recurrence rates (recurrence being defined as the development of a new sinus or abscess within the natal cleft occurring after wound healing had been achieved) between the NPWT and SWC Groups
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 1 month
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 3 months
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 6 months
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Scar assessment - using the Patient and Observer Scar Assessment Scale (POSAS) | 1 month
  The POSAS is made up of two scales: the patient scale and the observer scale; each of the six components is scored numerically on a scale of 1 to 10. The component scores are then added together; the worst scar would receive a score of 60, while the best scar would receive a score of 6
Scar assessment - using the Patient and Observer Scar Assessment Scale (POSAS) | 3 months
  The POSAS is made up of two scales: the patient scale and the observer scale; each of the six components is scored numerically on a scale of 1 to 10. The component scores are then added together; the worst scar would receive a score of 60, while the best scar would receive a score of 6
Scar assessment - using the Patient and Observer Scar Assessment Scale (POSAS) | 6 months
  The POSAS is made up of two scales: the patient scale and the observer scale; each of the six components is scored numerically on a scale of 1 to 10. The component scores are then added together; the worst scar would receive a score of 60, while the best scar would receive a score of 6
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 1 Month
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 3 Months
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 6 Months
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Health Economics evaluation of resource use and cost effectiveness using Negative Pressure Wound Therapy dressings | 6 Months
  Investigating resource use and cost effectiveness of single-use, prophylactic negative pressure wound therapy versus standard dressings for midline laparotomy wounds based on length of hospital stay and costs of dressings
Visual pain score questionnaire | Day of Surgery
  Measurement of pain intensity
Visual pain score questionnaire | 1 Month
  Measurement of pain intensity
Visual pain score questionnaire | 3 Months
  Measurement of pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Sean T Martin, Principal Investigator — St. James's Hospital, Ireland
Locations (10):
- Ireland (10):
  - Mayo University Hospital, Castlebar
  - University Hospital Cork, Cork
  - Beaumont Hospital, Dublin
  - St Michael's Hospital Dun Laoighre, Dublin
  - Tallaght University Hospital, Dublin
  - University Hospital Galway, Galway
  - St. Luke's Hospital, Kilkenny
  - University Hospital Limerick, Limerick
  - Midlands University Hospital, Tullamore
  - University Hospital Waterford, Waterford

IPD SHARING:
Plan to Share IPD: No